CLINICAL TRIAL: NCT02042625
Title: Optimal Positioning of Nasopharyngeal Temperature Probes: A Prospective Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 13-1443
Record Dates: First submitted 2013-12-06; First posted 2014-01-23 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nasopharyngeal (Other): The nasopharyngeal probe will be inserted into the nostril. The nasopharyngeal temperature will initially be recorded 45 minutes after anesthetic induction. The nasopharyngeal probe will then be withdrawn 2 cm and after a 3-minute equilibration period, nasopharyngeal temperatures will again be recorded. The nasopharyngeal probe withdrawal sequence will be repeated, 2 cm at a time, until only 2 cm remains in the nostril. There will be a total of 10 sets of nasopharyngeal temperatures obtained.
  Interventions: Procedure: Nasopharyngeal

INTERVENTIONS:
Procedure: Nasopharyngeal

SUMMARY:
Low body temperature (hypothermia) is often observed in anesthetized patients. Mild hypothermia increases complications such as surgical blood loss, postanesthesia recovery and the duration of hospitalization. To assess body temperature and minimize hypothermia-related complications, it is important to have accurate and reliable methods of measuring intraoperative core temperature. Common practice is to insert a nasopharyngeal (back of the throat from the nose) probe through one of the nostrils. However, there is no consensus or guideline regarding how deep the nasopharyngeal probe needs to be inserted. This study is being done to determine the insertion depth (or range of depths) that best approximates core temperature, which is temperature of the vital organs, e.g. heart, liver and lungs.

Participation in the trial will occur on the day of surgery. The subject will be asked to breathe through one nostril and then the other before receiving anesthesia. The less congested nostril will be selected for study. If there is no difference, then the investigator will use the right nostril.

Once under anesthesia, an esophageal temperature probe will be inserted to serve as a reference core temperature, which is used routinely in surgery. Then the nasopharyngeal probe will be inserted into the nostril.

Both nasopharyngeal and esophageal temperatures will initially be recorded 45 minutes after anesthetic induction. The nasopharyngeal probe will then be withdrawn 2 cm and after a 3-minute equilibration period, nasopharyngeal and esophageal temperatures will again be recorded. The nasopharyngeal probe withdrawal sequence will be repeated, 2 cm at a time, until only 2 cm remains in the nostril. There will be a total of 10 sets of nasopharyngeal and esophageal temperatures obtained.

ELIGIBILITY:
Inclusion Criteria:

* elective non-cardiac surgery scheduled to last at least 1.5 hours
* supine position anticipated
* general anesthesia with ETT

Exclusion Criteria:

* nasopharyngeal disease (e.g. sinusitis), upper airway abnormalities, or planned surgery in the region
* history of recent substantive epistaxis
* history of bleeding disorders
* therapeutic-dose anti-coagulation (aspirin and DVT prophylaxis permitted)
* contraindications to esophageal temperature probe insertion (e.g. known varices)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
insertion depth of nasopharyngeal probe for core temperature | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mi Wang, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States